CLINICAL TRIAL: NCT00502021
Title: Inflammatory Indicators and Arterial Stiffness in Patients With Severe Obesity. Response to Supplementation of Alpha Linolenic Acid
Brief Title: Use of Flaxseed(Alpha Linolenic Acid) Powder in Morbidly Obese Patients With Systemic Inflammation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Joel Faintuch, Associate Professor, Department of Gastroenterology, Sao Paulo University Medical School, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Flaxseed01
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Morbid Obesity; Atherosclerosis; Systemic Inflammation
Keywords: obesity; alpha linolenic acid; flaxseed; C-reactive protein; inflammation
MeSH Terms: conditions — Obesity, Morbid; Atherosclerosis; Obesity; Inflammation | interventions — Docosahexaenoic Acids; Linseed Oil; Fatty Acids, Omega-6

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Supplement of flaxseed powder (60 g/day)during 12 weeks
  Interventions: Dietary Supplement: Alpha-linolenic acid/ALA
- 2 (Placebo Comparator): Placebo powder supplement 60 g/day during 12 weeks
  Interventions: Dietary Supplement: Placebo
- 3 (Experimental): Flaxseed oil 30 ml/day (10 g ALA)during 12 weeks
  Interventions: Dietary Supplement: Alpha linolenic acid/ALA
- 4 (Placebo Comparator): Safflower oil 30 ml/day (no ALA) during 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Manioc powder (placebo) 60 g/day
  Other Names: Cassava powder
  Arms: 2
Dietary Supplement: Alpha-linolenic acid/ALA — Flaxseed powder 60 g/day (10 g ALA)
  Other Names: Linseed powder, omega- 3 fatty acid
  Arms: 1
Dietary Supplement: Alpha linolenic acid/ALA — Flaxseed oil 30 ml/day (10 g ALA)
  Other Names: Linseed oil, omega- 3 fatty acid
  Arms: 3
Dietary Supplement: Placebo — Safflower oil 30 ml/day
  Other Names: Omega 6 fatty acids
  Arms: 4

SUMMARY:
Preliminary studies have shown that flaxseed powder, rich in the omega-3 alpha-linolenic acid,is beneficial for the general inflammation present in morbidly obese subjects by decreasing elevated serum markers.As omega-3 fatty acids display additional properties including possible amelioration of atherosclerosis,a 3-month supplementation protocol was devised.Arterial stiffness and intima thickness will be measured in severely obese subjects, in order to document possible reduction of these variables as well.

DETAILED DESCRIPTION:
Population:Morbidly obese non-smoking patients of the Department of Gastroenterology, candidates for possible bariatric treatment Criteria for inclusion: Males and females, 18- 65 years old, body mass index/BMI > 40 kg/m2 (or > 35 kg/m2 with comorbidities), non-hospitalized and receiving general oral diet, with elevated C-reactive protein/ CRP (> 5mg/L), and signing informed consent; Criteria for exclusion: SIRS, shock, coma or organ failure, fever or infectious foci, cancer with or without chemo/radiotherapy, inflammatory illnesses (rhematic, gastrointestinal or other), transplantation or immunologic diseases, trauma, surgery or hospitalization in the last 30 days, use of steroidal or non-steroidal anti-inflammatory or immune-modulating agents or antibiotics, and refusal to participate in the study; Dietetic routine: Daily flaxseed powder (Farinha de linhaca dourada) 60 g/day (232 kcal , containing 10 g of alpha-linolenic acid/ALA) or placebo (commercial manioc flour 60 g/day, 120 kcal)) during 12 weeks. An additional 60 subjects (30 patients, 30 controls) will ve managed with 30 ml/day flaxseed oil (10 g of alpha-linolenic acid/ALA) or 30 ml/day placebo (safflower oil).

Methods: Clinical questionnaire,nutritional assessment(Weight, height, BMI) Biochemical tests: Hemoglobin (HB) , white blood cell count (WBC), total cholesterol (CHOL) and fractions (HDL, LDL, VLDL), triglycerides (TRIG), blood glucose (GLU), serum albumin (ALB),insulin (INS), leptin (LEP),C-reactive protein (CRP), serum amyloid A (SAA), complement fractions C3 and C4, coagulation profile Atherosclerosis markers: Arterial stiffness (aorta) and intima thickness (common carotid artery)

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* 18- 65 years old
* Body mass index/BMI > 40 kg/m2 (or > 35 kg/m2 with comorbidities)
* Non-hospitalized and receiving general oral diet
* With elevated C-reactive protein/ CRP (> 5mg/L); and
* Signing informed consent

Exclusion Criteria:

* SIRS, shock, coma or organ failure,
* Fever or infectious foci
* Cancer with or without chemo/radiotherapy
* Inflammatory illnesses (rhematic, gastrointestinal or other), transplantation or immunologic diseases
* Trauma, surgery or hospitalization in the last 30 days
* Use of steroidal or non-steroidal anti-inflammatory or immune-modulating agents or antibiotics; and
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in arterial stiffness/intima thickness | 12 weeks

SECONDARY OUTCOMES:
Improvement in inflammatory markers and serum lipids | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joel Faintuch, MD,PhD, Study Chair — Sao Paulo University Medical School; Patricia C Marques, MD, Principal Investigator — Hospital das Clinicas
Locations (1):
- Hospital das Clinicas-ICHC-9th Floor- Av. Eneias C. Aguiar 255, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Faintuch J, Horie LM, Barbeiro HV, Barbeiro DF, Soriano FG, Ishida RK, Cecconello I. Systemic inflammation in morbidly obese subjects: response to oral supplementation with alpha-linolenic acid. Obes Surg. 2007 Mar;17(3):341-7. doi: 10.1007/s11695-007-9062-x. PMID 17546842
- [Background] Faintuch J, Horie LM, Schmidt VD, Barbeiro HV, Barbeiro DF, Soriano FG, Cecconello I. Obesity, inflammation, vascular reactivity, and cardiocirculatory events. Clinics (Sao Paulo). 2007 Jun;62(3):357-8. doi: 10.1590/s1807-59322007000300023. No abstract available. PMID 17589679